CLINICAL TRIAL: NCT01109264
Title: Study of Bendamustine Hydrochloride Injection in Previously Untreated Chronic Lymphocytic Leukemia Patients
Brief Title: Bendamustine Hydrochloride Injection for Initial Treatment of Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIM-79-001
Record Dates: First submitted 2010-04-19; First posted 2010-04-23 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Bendamustine Hydrochloride; Chlorambucil
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Chlorambucil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bendamustine Hydrochloride (Experimental)
  Interventions: Drug: Bendamustine hydrochloride injection
- Chlorambucil (Active Comparator)
  Interventions: Drug: Chlorambucil

INTERVENTIONS:
Drug: Bendamustine hydrochloride injection — d1-2, i.v.gtt, 100mg/m2, 28 days per cycle, at most 6 cycles
  Arms: Bendamustine Hydrochloride
Drug: Chlorambucil — d1-d2, d15-d16, p.o., 0.4mg/kg/day, 28 days per cycle, at most 6 cycles
  Arms: Chlorambucil

SUMMARY:
To compare the clinical efficacy and safety of bendamustine hydrochloride versus chlorambucil for initial treatment of chronic lymphocytic leukemia

DETAILED DESCRIPTION:
Patients will be assessed for response after three cycles of treatment. Two additional cycles are recommended for CR, PR or SD patients, up to a maximum limit of six cycles in total. Patients will be followed up every three months until disease progression or death.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of CLL according to National Cancer Institute (NCI) Working Group criteria
* No prior treatment for CLL
* Binet stage B or C
* ECOG performance status ≤ 2
* Life expectancy ≥3 months
* AST and ALT ≤ 3 x ULN; Total bilirubin ≤ 2 x ULN; Creatinine clearance ≥ 40 mL/min
* Written informed consent

Exclusion Criteria:

* Patients were diagnosed with or treated for malignant tumors other than CLL (including central nervous system lymphoma) within one year prior to entering the study
* Transformation to Richter's syndrome, or prolymphocytic leukemia (PLL)
* Autoimmune hemolytic anemia requiring glucocorticoid therapy
* Autoimmune thrombocytopenia requiring glucocorticoid therapy
* Participation in any other clinical trials within 4 weeks prior to study entry
* Any of the following conditions: severe heart failure; cardiomyopathy; myocardial infarction within 6 months; severe, uncontrolled diabetes; severe, uncontrolled hypertension; active, uncontrolled infection; central nervous system dysfunction
* Patients received major surgery within 30 days prior to study entry
* Pregnant or lactating women
* Allergic to study drug or mannitol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2010-03; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | after 3 cycles and 6 cycles

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | December 2013
Duration of Remission (DR) | December 2013
Overall Survival (OS) | December 2013
The incidence and severity of adverse events | Up to 2 years after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiang Shen, Dr., Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Affiliated to Shanghai JiaoTong University School of Medicine, Shanghai, China